CLINICAL TRIAL: NCT06392711
Title: UW23129: A Phase I Dose-Escalation Trial of Mesenchymal Stromal Cells in Patients With Medical Xerostomia
Brief Title: Dose-Escalation Trial of Mesenchymal Stromal Cells in Patients With Medical Xerostomia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0386; A534290 (Other: UW- Madison); SMPH/MEDICINE/RHEUMATOL (Other: UW- Madison); UW23129 (Other: UW- Madison); Protocol Version 11/29/25 (Other: UW- Madison)
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-10

CONDITIONS: Xerostomia; Graft-versus-host-disease; Sjogren's Disease
MeSH Terms: conditions — Xerostomia; Graft vs Host Disease; Sjogren's Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MSCs Dose Level 0 into one submandibular gland (Active Comparator): 6 subjects will receive Mesenchymal Stromal Cells (MSC) at Dose Level 0, which is 10 (8-12) x10^6 MSCs in a single submandibular gland. If this dose is deemed tolerable when injected into a single submandibular gland, this dose will be administered to both submandibular glands in the initial subjects in the dose escalation arm.
  Interventions: Biological: Mesenchymal Stromal Cells (MSC) Dose Level 0
- MSCs into both submandibular glands - Dose Escalation Cohort (Active Comparator): 8-18 subjects in the Dose Escalation phase of study will receive MSCs into both submandibular glands. The initial subjects in this cohort will receive Dose Level 0: 10 (8-12) x10^6 MSCs/gland. If this dose is tolerated, subsequent subjects will receive Dose Level 1: 20 (16-24) x10^6 MSCs/gland. The highest tolerated dose (recommended phase II dose or RP2D) will be administered to the subjects in the Expansion Cohort.
  Interventions: Biological: Mesenchymal Stromal Cells (MSC) Dose Level 0; Biological: Mesenchymal Stromal Cells (MSC) Dose Level 1
- MSCs into both submandibular glands - Expansion Cohort (Active Comparator): 12 subjects in Expansion Cohort will receive MSCs into both submandibular glands at the RP2D.
  Interventions: Biological: Mesenchymal Stromal Cells (MSC) Dose Level 0; Biological: Mesenchymal Stromal Cells (MSC) Dose Level 1

INTERVENTIONS:
Biological: Mesenchymal Stromal Cells (MSC) Dose Level 0 — 10 (8-12) x 10^6 MSCs
Biological: Mesenchymal Stromal Cells (MSC) Dose Level 1 — 20 (16-24) x 10^6
  Arms: MSCs into both submandibular glands - Dose Escalation Cohort; MSCs into both submandibular glands - Expansion Cohort

SUMMARY:
The goal of this clinical trial is to evaluate the safety and tolerability of injecting certain cells produced in bone marrow called mesenchymal stromal cells (MSCs) into salivary glands. The main question it aims to answer is whether injection of MSCs into salivary glands results in any improvement in dry mouth.

Participants will:

* have bone marrow collected using a needle
* undergo a salivary gland ultrasound
* complete questionnaires
* receive an injection of the bone marrow cells into a salivary gland

DETAILED DESCRIPTION:
This single-center phase I dose-escalation with expansion cohort, open label, non-randomized, non-placebo controlled, single group assignment study will assess the safety and tolerability of mesenchymal stromal cells (MSCs) for treatment of xerostomia, focusing on xerostomia with inflammatory etiology (e.g., Sjögren's disease [SjD], graft-versus-host disease [GVHD]). An initial cohort of subjects (n=6) will receive a unilateral injection of MSCs at dose level 0. If unilateral treatment is tolerated, a dose escalation cohort (n=8-18) will receive bilateral injection of MSCs. Dose escalation will proceed using a standard 3+3 design and once the recommended phase II dose (RP2D) is defined, 12 additional patients will be accrued to the expansion phase.

Following the completion of screening/baseline procedures, eligible participants will undergo bone marrow aspiration in order to obtain MSCs.

The MSC investigational product will be injected into one or both submandibular glands under local anesthesia at the interventional visit.

ELIGIBILITY:
Inclusion Criteria:

* Xerostomia, defined as an unstimulated salivary flow <1.2 mL in 5 minutes documented at any time following xerostomia diagnosis and prior to enrollment
* Xerostomia not resulting from radiotherapy (medical xerostomia)
* ≥ 18 years of age, ≤ 90 years of age
* Karnofsky performance status ≥ 70, patient eligible for bone marrow aspirate with wakeful anesthesia
* Willing and able to give informed consent
* Radiographically confirmed bilateral submandibular glands
* If female of childbearing potential, negative pregnancy test
* Males and females of childbearing potential willing to use acceptable contraception
* Laboratory Values (within 28 calendar days of enrollment):

  * Hgb ≥ 9 g/dL (5.58 mmol/L)
  * Platelets ≥ 100,000/µL
  * ANC ≥ 1000/µL
  * Lymphocytes ≥ 800/µL
  * PT/INR and PTT within normal limits based on age/sex

Exclusion Criteria:

* Patients with one submandibular gland
* Sialolithiasis
* Poorly-controlled diabetes mellitus (HbA1c ≥ 7%)
* Patients who initiated any diuretic therapy before developing dry mouth symptoms and are still on diuretic therapy and the referring provider believes the dryness symptoms are driven by diuretic use
* Untreated oral candidiasis based on physical exam at enrollment
* Malignancy within the last 2 years (except adequately treated stage I lung cancer, low risk prostate cancer that has been treated or is undergoing active surveillance, adequately treated non-melanoma skin cancer, adequately treated DCIS, or adequately treated stage I cervical cancer)
* For patients on immunosuppressive therapy, must be on stable dose of immunosuppressive therapy for at least 2 months, allowing for dose adjustments for blood levels of drugs
* Transfusion dependency
* Life expectancy ≤ 6 months as determined by the investigator
* Use of investigational drugs, biologics, or devices within 30 calendar days prior to enrollment
* Pregnant or lactating women or those who plan to become pregnant during the study
* Not suitable for study participation due to other reasons at discretion of investigators.
* Enrollment in another clinical study possibly interfering with the endpoints of this study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants experiencing DLT of submandibular pain | 1 month post-injection
  Recommended phase II dose (RP2D) will be determined by the proportion of subjects experiencing the dose-limiting toxicity (DLT) of submandibular pain > 5 on a standard 10-point pain scale of 0-10 at 1-month after MSC injection
Proportion of participants experiencing DLT as serious adverse events (AEs) | 1 month post-injection
  RP2D will be determined by the proportion of subjects experiencing the dose-limiting toxicity (DLT) of any serious AE within one-month post-injection
Proportion of participants experiencing DLT as pre-specified toxicities | 1 month post-injection
  RP2D will be determined by the proportion of subjects experiencing the dose-limiting toxicity (DLT) of any selected toxicity that is specified in the protocol within one-month post-injection

SECONDARY OUTCOMES:
Change in xerostomia scores | Baseline to 24 months
  Xerostomia will be assessed by quality of life xerostomia (XeQoL) scores. XeQoL is a 15-item questionnaire, where items 1-14 are scored as: 0=not at all; 1=a little; 2=somewhat; 3=quite a bit; 4=very much. Item 15 is scored as: 0=delighted; 1=mostly satisfied; 2=mixed: equally satisfied/dissatisfied; 3= mostly dissatisfied; 4=terrible. Lower scores indicate less impact of mouth/throat dryness on QoL, and higher scores indicate great impact on QoL.
Change in salivary function-rate of salivary production | Baseline, 1 month, 3 months, 6 months, 12 months, and 24 months
  Salivary function determined by measurement of salivary production (g/5 minutes); Unstimulated saliva production will be measured by participants allowing saliva to pool in the mouth over a 5 minute period, then gently guiding saliva into a saliva collection aid; Simulated saliva production will be measured by participants chewing inert gum base to the pace of a metronome (70 beats/minute) while expectorating saliva into a saliva collection aid for 5 minutes. Cryovials containing saliva will be weighed before and after saliva collection and the difference in weight (g) will represent the amount of saliva produced in 5 minutes for each condition.
Change in salivary function-saliva composition | Baseline, 1 month, 3 months, 6 months, 12 months, and 24 months
  Salivary function determined by compositional analysis of saliva sample - amylase (mU/mL). Low in disease, hypothesized to increase with intervention.
Change in salivary function-saliva composition | Baseline, 1 month, 3 months, 6 months, 12 months, and 24 months
  Salivary function determined by compositional analysis of saliva sample - mucins (MUC5B in mU/mL) assessed using ELISA. Low in disease, hypothesized to increase with intervention.
Change in salivary function-saliva composition | Baseline, 1 month, 3 months, 6 months, 12 months, and 24 months
  Salivary function determined by compositional analysis of saliva sample; pH assessed using pH meter. Low in disease, hypothesized to increase with intervention.
Change in salivary function-saliva composition | Baseline, 1 month, 3 months, 6 months, 12 months, and 24 months
  Salivary function determined by compositional analysis of saliva sample - total protein (mg/mL). High levels in disease, hypothesized to decrease with intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sara McCoy, MD, PhD, Principal Investigator — University of Wisconsin, Madison; Jacques Galipeau, MD, Study Director — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No